CLINICAL TRIAL: NCT01191970
Title: Investigating Potential Determinants of Breast-Feeding Probability: Epidural Analgesia, Beta-Endorphin Concentrations in Colostrum, and Infant Feeding Behavior
Brief Title: Epidural Analgesia, Beta-Endorphin Concentrations in Colostrum, and Infant Neurobehavior as Breast-Feeding Predictors
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn from IRB
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Charles Smith, M.D., MetroHealth Medical Center
Other Study IDs: 1-Szabo
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Breastfeeding; Lactation; Analgesia
Keywords: epidural; beta-endorphins; breast-feeding; colostrum; feeding
MeSH Terms: conditions — Breast Feeding; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Colostrum samples collected 2x/d for duration of postpartum hospital stay, which is, on average, 2d.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epidural recipients: Subjects who received epidural analgesia during labor
- Non-epidural recipients: Subjects who did not receive epidural analgesia during labor

SUMMARY:
Presently, the literature addressing the relationship between epidural analgesia and likelihood of breast-feeding is inconclusive. Numerous studies have found that epidurals, administered prior to vaginal delivery of a full-term, healthy neonate, significantly decrease lactation success at follow-up times ranging from 24 hours to 6 months postpartum. One proposed mechanism is that analgesics, by decreasing maternal pain during labor, decrease maternal endorphin production and result in the transmission of lower endorphin levels to the neonate during breast-feeding. Lower endorphin levels, in turn, may render the neonate less likely to suckle optimally. Other studies have found that epidural analgesia does not significantly decrease lactation success when used during the vaginal delivery of a full-term, healthy neonate.

Although most studies to date have compared the breast-feeding success of epidural recipients and non-recipients at various points postpartum, they do not specifically note whether deficient feeding behaviors on the part of the infant contribute to failed breast-feeding. The present study uses the LATCH assessment tool to score the infant's ability to latch onto the breast and the presence of audible swallowing, as well as the mother's level of physical comfort with breast feeding, whether she can successfully position the infant for feeding on her own, and whether her nipples are inverted, everted, or flat. Thus, the LATCH assessment enables the separation of multiple factors that may contribute to breast-feeding failure. A multivariate regression analysis will determine how strongly the probability of breast-feeding at hospital discharge correlates with epidural duration, LATCH scores, and beta-endorphin concentrations in colostrum.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Vaginal delivery of a single live neonate at MetroHealth Medical Center's Main Campus

Exclusion Criteria:

* Delivery by Caesarean section
* Admission to the NICU following delivery
* Neonatal or maternal pathologies that would obviously impede normal breast-feeding activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is open to all women, aged 18 and over, who are inpatients on the postpartum floor of MetroHealth Medical Center following the vaginal delivery of a single, healthy neonate. A neonate is "healthy" if neither of the following two conditions exists: 1) admission to the neonatal intensive care unit (NICU) following delivery and 2) pathologies, in either mother or baby, that would be reasonably expected to impede normal breast-feeding activity.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Breast-Feeding at Discharge | Entire duration of postpartum hospital stay, average 2 days
  The primary outcome measure is whether the subject is breast-feeding her infant, either exclusively or with bottle supplementation, at the time of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Smith, M.D., Study Director — Dept. of Anesthesiology, MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Baumgarder DJ, Muehl P, Fischer M, Pribbenow B. Effect of labor epidural anesthesia on breast-feeding of healthy full-term newborns delivered vaginally. J Am Board Fam Pract. 2003 Jan-Feb;16(1):7-13. doi: 10.3122/jabfm.16.1.7. PMID 12583645
- [Background] Beilin Y, Bodian CA, Weiser J, Hossain S, Arnold I, Feierman DE, Martin G, Holzman I. Effect of labor epidural analgesia with and without fentanyl on infant breast-feeding: a prospective, randomized, double-blind study. Anesthesiology. 2005 Dec;103(6):1211-7. doi: 10.1097/00000542-200512000-00016. PMID 16306734
- [Background] Chang ZM, Heaman MI. Epidural analgesia during labor and delivery: effects on the initiation and continuation of effective breastfeeding. J Hum Lact. 2005 Aug;21(3):305-14; quiz 315-9, 326. doi: 10.1177/0890334405277604. PMID 16113019
- [Background] Henderson JJ, Dickinson JE, Evans SF, McDonald SJ, Paech MJ. Impact of intrapartum epidural analgesia on breast-feeding duration. Aust N Z J Obstet Gynaecol. 2003 Oct;43(5):372-7. doi: 10.1046/j.0004-8666.2003.t01-1-00117.x. PMID 14717315
- [Background] Zanardo V, Nicolussi S, Carlo G, Marzari F, Faggian D, Favaro F, Plebani M. Beta endorphin concentrations in human milk. J Pediatr Gastroenterol Nutr. 2001 Aug;33(2):160-4. doi: 10.1097/00005176-200108000-00012. PMID 11568517
- [Background] Kumar SP, Mooney R, Wieser LJ, Havstad S. The LATCH scoring system and prediction of breastfeeding duration. J Hum Lact. 2006 Nov;22(4):391-7. doi: 10.1177/0890334406293161. PMID 17062784
- [Background] Volmanen P, Valanne J, Alahuhta S. Breast-feeding problems after epidural analgesia for labour: a retrospective cohort study of pain, obstetrical procedures and breast-feeding practices. Int J Obstet Anesth. 2004 Jan;13(1):25-9. doi: 10.1016/S0959-289X(03)00104-3. PMID 15321436
- [Background] Gray L, Miller LW, Philipp BL, Blass EM. Breastfeeding is analgesic in healthy newborns. Pediatrics. 2002 Apr;109(4):590-3. doi: 10.1542/peds.109.4.590. PMID 11927701